CLINICAL TRIAL: NCT03077893
Title: A Multi-Center, Sham-Controlled, Double-Blind Randomized Withdrawal Study of PEMF Therapy to Evaluate Vibration Perception Threshold and Thermal Sensory in Subjects With Diabetic Peripheral Neuropathy in the Lower Extremity
Brief Title: Study of PEMF to Evaluate VPT and Thermal Sensory in Subjects With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBI.2017.001
Record Dates: First submitted 2017-02-28; First posted 2017-03-13 (Actual); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: Subjects deemed "responders" after active treatment will be randomized in a 1:1 ratio to either active treatment or a sham device.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham devices will look identical to active devices. This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Group (Experimental): Treatment with active Provant Therapy System
  Interventions: Device: Active Provant Therapy System
- Sham Group (Sham Comparator): Treatment with Inactive (sham) Provant Therapy System
  Interventions: Device: Inactive (sham) Provant Therapy System

INTERVENTIONS:
Device: Active Provant Therapy System — Treatment with active Provant Therapy System
  Arms: Active Group
Device: Inactive (sham) Provant Therapy System — Treatment with Inactive (sham) Provant Therapy System
  Arms: Sham Group

SUMMARY:
A study to demonstrate the effectiveness of PEMF treatment compared to sham treatment in changing Vibration Perception Threshold (VPT) and Thermal Sensory (QST) in patients with diabetic peripheral neuropathy (DPN) when treatment is administered twice daily through 120-day period.

DETAILED DESCRIPTION:
Multi-center, sham-controlled, double-blind, enriched enrollment, randomized withdrawal clinical trial conducted on subjects with bilateral symmetrical diabetic peripheral neuropathy. Eligible subjects will include those between 22 and 80 years of age with Type 1 or Type 2 diabetes having persistent pain, numbness, tingling, or burning in both feet despite treatment. Eligible subjects will receive two active treatment devices (one for each foot, to allow simultaneous treatment) and treat at home, twice daily for 60 days after which they will return to the clinic at Day 61 for a response assessment. Subjects that are determined to be responders at Day 61 (subjects that achieve a 1-point decrease in the average pain score over the last 24 hours using the Numeric Pain Rating Scale (NPRS)) will be randomized 1:1 to either active treatment or inactive sham devices and will continue treating through Day 120. Subjects that are determined to be non-responders at Day 61 will continue treating with the active devices given at enrollment and will return to the clinic at Day 75 and Day 91 for a response assessment. If a subject is determined to be a responder at Day 75, they will be randomized 1:1 to receive either active treatment or inactive sham and will continue treating through Day 120. If a subject is determined to be a responder at Day 91, they will be randomized 1:1 to receive either active treatment or sham and will continue to treat through Day 120. If a subject continues to be a non-responder at Day 91 they will be terminated from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater than or equal to 22 years and less than 80 years of age.
2. Subject has documented Type 1 or Type 2 diabetes mellitus (receiving insulin, diet controlled, or taking parenteral hypoglycemic agents)
3. Subject is on a stable antidiabetic regimen (medication and/or diet) to control their diabetes for at least 30 days prior to Screening.
4. Subject has an HbA1c <10% at Screening or within 2 months of Screening.
5. Subject has daily pain attributed to bilateral symmetrical Diabetic Peripheral Neuropathy with numbness, tingling, and/or burning based on clinical judgement for at least 6 months prior to screening.
6. Subject's pain or discomfort from DPN is identifiable.
7. Subject is in pain Phase 2, 3, or 4 as per the Phasing of Neuropathy Scale.
8. Subjects average pain over the last 24 hours is ≥3 based on the 11-point Numeric Pain Rating Scale (NPRS) at the Screening Visit.
9. Subject has adequate lower extremity pulse in both feet and no intermittent claudication.
10. Subject is able to ambulate independently without assistive devices.
11. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol.
12. Female subjects must be post-menopausal, surgically sterile, abstinent, or practicing (or agrees to practice) an effective method of birth control if they are sexually active for the duration of the study (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Exclusion Criteria:

1. Subject is in pain Phase 1 or 5 as per the Phasing of Neuropathy Scale.
2. Subject has an active, open ulcer on the lower extremities.
3. Subject has peripheral vascular disease defined as absence of more than one foot pulse per foot and/or ABI <0.8 and >1.4 and/or history of angioplasty or peripheral bypass surgery within 6 months of the Screening Visit.
4. Subject has venous insufficiency as classified by the Venous Insufficiency Classification System of grade C6.
5. Subject has undergone nerve decompression surgery on the lower extremities.
6. Subject has a history of previous kidney, pancreas, cardiac transplantation, or severe renal disease.
7. Subject has been diagnosed with non-diabetic chronic inflammatory neuropathic disease (e.g. end stage renal disease, hepatitis C, chemotherapy induced neuropathy, known connective tissue disease, systemic lupus).
8. Subject has peripheral vascular disease requiring revascularization of lower limb or amputation or evidence of ulcer amputation.
9. Subject has clinically significant cardiovascular disease within 6 months prior to screening (unstable or poorly controlled hypertension, transient ischemic attack, MI, unstable angina, arrhythmia, any heart surgery, stent placement, heart disease).
10. Subject has a history of any uncontrolled medical illness that in the Investigators judgment places the subject at unacceptable risk for receipt of PEMF therapy.
11. Subject requires or anticipates the need for surgery of any type or travel during the treatment period.
12. Subject has a total foot depth (most inferior aspect of the medial malleolus to the plantar aspect of the foot when residing on a treatment pad) of >8 cm.
13. Subject has received any investigational drug or device within 30 days prior to the Screening Visit or within 6 weeks prior to the Screening Visit for long acting lidocaine injection products.
14. Subject has used systemic corticosteroids within 3 months of the Screening Visit.
15. Subject has a history of malignancy within the past 5 years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area and/or localized in situ carcinoma of the cervix.
16. Subject has a serious psychosocial co-morbidity.
17. Subject has a history of drug or alcohol abuse, as confirmed by urine drug screen, within one year prior to the Screening Visit.
18. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
19. Subject is currently pregnant or planning on becoming pregnant prior to Day 121.
20. Subject has previously treated with PROVANT® Therapy System within 60 days on the lower extremity.
21. Subject is unwilling or unable to follow study instructions or comply with the treatment regimen, diary documentation, and study visits.
22. Subject has pain from any other source that can confuse the assessment of the pain associated with DPN.
23. Subject has a clinically significant foot deformity (Charcot's syndrome or club foot).
24. Subject has received nerve blocks for neuropathic pain within 4 weeks of the Screening Visit.
25. Subject has been diagnosed with mononeuropathy.
26. Subject has a skin condition that could alter their sensation.
27. Subject has had a previous surgery to the spine or lower extremity with residual symptoms of pain or difficulty with movement.
28. Subject has moderate or severe arthropathy (RA, OA, Gout) that causes discomfort during casual walking or stair climbing.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Tallas, DPM, Principal Investigator — Associated Foot & Ankle Specialists, LLC
Locations (1):
- Associated Foot & Ankle Specialists, LLC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 44 subjects were enrolled into the trial and given active Provant Therapy. A total of 7 subjects dropped out of the study prior to being randomized 1:1 active to sham. Since these subjects withdrew from the study prior to assignment to an arm, they are not included in the randomized total of 37 (18 active and 19 sham).
Period: Overall Study
Arm/Group | Active Group | Sham Group
Started | 18 | 19
Completed | 14 | 16
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Sham Group | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 62.5 [39 to 86] | 62.05 [36 to 76] | 62.27 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 15 | 16 | 31
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Vibration Perception Threshold (VPT)
Description: A non-invasive test used in quantifying sensation/sensitivity to vibration in evaluating sensory dysfunction associated with diabetic neuropathy
Time Frame: Baseline to End of Treatment (Day 121)
Measure: Mean (Standard Deviation); unit: amplitude in microns
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 17 | 18
amplitude in microns
  Big Toe, change in VPT | 9.26 (32.67) | -3.59 (21.08)
  Plantar Aspect, change in VPT | 9.18 (32.10) | 1.184 (19.66)

2. Primary Outcome: Quantitative Sensory Testing (QST)
Description: QST is a noninvasive test used in peripheral nervous system disorders for thermal sensory testing.
Time Frame: Baseline to End of Treatment (Day 121)
Population: Number analyzed in outcome measure table is less than overall number analyzed due to drop-outs and technical issues with the QST machine.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 18 | 19
Participants
  Baseline QST, Abnormal Result: number analyzed (Participants) | 15 | 14
  Baseline QST, Abnormal Result | 9 | 8
  Baseline QST, Normal Result: number analyzed (Participants) | 15 | 14
  Baseline QST, Normal Result | 6 | 6
  Day 121 QST, Abnormal Result: number analyzed (Participants) | 11 | 12
  Day 121 QST, Abnormal Result | 4 | 4
  DAy 121 QST, Normal: number analyzed (Participants) | 11 | 12
  DAy 121 QST, Normal | 7 | 8

3. Secondary Outcome: Nerve Conduction Velocity (NCV) - Velocity
Description: NC-stat® DPNCheck® will be used to record NCV at Baseline and Day 121. Outcome Measure Data table displays change in NCV from Baseline to Day 121.
Time Frame: The sural nerve conduction velocity will be recorded at the Enrollment Visit and end of study visit (Day 121).
Measure: Mean (Standard Deviation); unit: micro volts
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 16 | 13
micro volts | 1.69 (15.15) | -4.23 (13.49)

4. Secondary Outcome: Skin Perfusion Pressures (SPP)
Description: The Vasamed Sensilase PAD-IQ will be used to record SPP. This machine measures pressure (in mm Hg) of microcirculation using a laser Doppler sensor. Outcome Measure Data Table below displays change from Baseline to Day 121.
Time Frame: SPP will be conducted at the Enrollment Visit, Day 61, and end of study visit (Day 121).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 17 | 15
mmHg
  Change in Dorsal SPP | .35 (34.54) | 3.07 (40.16)
  Change in Medial Plantar SPP | -12.11 (32.98) | -2.06 (32.38)

5. Secondary Outcome: Pain Intensity (PI)
Description: Mean change from Baseline to Day 121, using a validated 11-point Numeric Pain Rating Scale (NPRS) with scores 0-10, where 0 = no pain and 10 = worst possible pain.
Time Frame: Collected as patient-reported outcomes on a paper diary and at the Enrollment visit to obtain a baseline value and on Days 61, 75, and 91
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 13 | 15
units on a scale | -2.69 (2.47) | -2.04 (2.67)

6. Secondary Outcome: Brief Pain Inventory (BPI); Question on Pain Right Now.
Description: The BPI long form will be administered at the Enrollment Visit, Day 30, 61, 91, and end of study visit (Day 121). Results for question #15 on Pain Right Now displayed below. Subject were asked to rate pain right now on a scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Change in BPI, pain right now question, from Baseline to Day 121.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 17 | 17
units on a scale | -1.65 (3.02) | -1.71 (2.78)

7. Secondary Outcome: Brief Fatigue Inventory (BFI)
Description: A 4-question assessment that assesses the level of fatigue and the impact of the fatigue on daily function over the last 24 hours. BFI is patient reported and collected at the Enrollment Visit, Days 30, 61, 91, and end of study visit (Day 121). A global fatigue score was calculated by averaging all of the values on the questionnaire and results for the change from Baseline to Day 121 are displayed below. The scale ranged from 0 (no fatigue/does not interfere) to 10 (as bad as you can imagine/completely interferes).
Time Frame: Change from Baseline to Day 121 in BFI.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 17 | 18
units on a scale | -1.65 (3.13) | -2.3 (1.98)

8. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: A 7-choice validated categorical scale of overall change in status since initiation of treatment with the study device.PGIC was collected every 7 days in the paper diary, immediately following the morning treatment. Subjects were asked: Since the start of the study, my overall status is? Choices on the scale included: Very much worse, much worse, minimally worse, no change, minimally improved, much improved and very much improved.
Time Frame: PGIC results at Day 121 displayed below.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 18 | 19
Participants
  Not Reported | 8 | 5
  Very Much Worse | 1 | 1
  Much Worse | 1 | 2
  Worse | 5 | 1
  Improved | 1 | 2
  Very Improved | 0 | 1
  Very Much Improved | 0 | 3
  No Change | 2 | 4

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: A patient reported 14 question assessment that detects the status of depression and anxiety. Subjects completed the assessment at the Enrollment Visit, Days 30, 61, 91, and end of study visit (Day 121). The total score for anxiety and the total score for depression was calculated at Day 121. Low scores represent normal (0-7) while high scores represent abnormal (11-21).
Time Frame: Change in Depression and Anxiety from Baseline to Day 121.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 17 | 18
units on a scale
  Mean change in depression | -.08 (2.23) | -.50 (2.81)
  Mean change in anxiety | -.12 (2.55) | -.94 (4.53)

10. Secondary Outcome: Neuro-QoL
Description: A validated set of health-related quality of life measures that are domain specific.Subjects will completed 6 domains: (1) Pain, (2) Lost/Reduced Feeling, (3) Diffuse Sensory Motor Symptoms, (4) Restrictions in Activities of Daily Living, (5) Disruptions in Social Relationships, and (6) Emotional Distress.The short forms were completed by the subject at the Enrollment Visit and end of study visit (Day 121). Each question in the domain was rated on a symptom scale from 1 (never) to 5 (all the time) and a bothersome scale from 1 (none) to 3 (very much).
  The total score for the domain was calculated by multiplying the symptom score by the bothersome score. The scale range is from 1 to 15 where the minimum (best/least symptomatic) score is 1 and the maximum (worst/most symptomatic) score is 15.
Time Frame: Change in each domain from Baseline to Day 121 is displayed below.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 16 | 17
units on a scale
  Change in Domain 1: Pain | -.22 (.84) | -.54 (.90)
  Change in Domain 2: Lost/Reducsed Feeling | -.02 (1.13) | -.37 (.97)
  Change in Domain 3: Diffuse Sensory Motor Symptoms | .06 (.52) | -.35 (.80)
  Change in Domain 4: Restrictions in Activities | -.12 (1.41) | -.5 (1.16)
  Change in Domain 5: Disruptions | -.13 (.45) | -.15 (.84)
  Change in Domain 6: Emotional Distress | -.25 (.52) | -.29 (1.07)

11. Secondary Outcome: Nerve Conduction Velocity (NCV) - Amplitude
Description: as for outcome 3
Time Frame: The sural nerve conduction amplitude will be recorded at the Enrollment Visit and end of study visit (Day 121).
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 16 | 13
meters/second | 1.56 (7.68) | 4.38 (13.21)

ADVERSE EVENTS:
Time Frame: Adverse events were collected and recorded for approximately 9 months, from 16 March 2017 to 21 December 2017. Adverse Events are separated out between the "2 month lead-in active", "sham group" and "active group".
Description: Definition does not differ.
Groups:
- 2 Month Lead-in Active Group: Treatment with active Provant Therapy System. Subjects treated with active device during the lead-in part of the study (prior to randomization).
- Active Group: Subjects randomized to treat with active Provant Therapy System.
- Sham Group: Subjects randomized to treat with sham device.
Arm/Group | 2 Month Lead-in Active Group | Active Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 8/44 | 3/44 | 2/44
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 2/44 | 0/44 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Month Lead-in Active Group (N=44) | Active Group (N=44) | Sham Group (N=44)
Elevated troponins and shortness of breath (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Concussion / Cerebrovascular Accident (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Month Lead-in Active Group (N=44) | Active Group (N=44) | Sham Group (N=44)
Pain in feet/foot (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated or arising from the performance of this Agreement is not permitted without the prior written consent of Regenesis. Such consent may be contingent on Regenesis' review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03077893/Prot_SAP_000.pdf